CLINICAL TRIAL: NCT02737878
Title: Reshaping the Path of Mild Cognitive Impairment by Refining Exercise Prescription: Understanding Training Type and Exploring Mechanisms
Brief Title: Reshaping the Path of Mild Cognitive Impairment by Refining Exercise Prescription
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of British Columbia (Other)
Responsible Party: Principal Investigator, Teresa Liu-Ambrose, Principal Investigator, University of British Columbia
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Treatment
Other Study IDs: H15-02181
Record Dates: First submitted 2016-04-11; First posted 2016-04-14 (Estimated); Last update posted 2026-01-13 (Actual); Status verified 2026-01

CONDITIONS: Mild Cognitive Impairment
MeSH Terms: conditions — Cognitive Dysfunction | interventions — Resistance Training

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Aerobic Training and Resistance Training (AT&RT) (Experimental): The AT&RT program will be a four-times-per week program. Twice a week will be aerobic training (AT) with a series of standardized AT exercise stations. Participants rotate through each station within the 40-min training duration with approx. 1-min rest between stations. Participants will exercise initially at approximately 50% of their age specific target heart rate reserve and gradually progress to reach the target of 80% of HRR. The other two days a week will be resistance training (RT) in which a pressurized air system and free weights will be used to provide the training stimulus. The initial intensity of the training stimulus will be set to a weight where participants can complete 2 sets of 10-15 repetitions. Training intensity will then progress on a cyclic basis from 45 to 85% of predicted 1 repetition maximum (1RM) as determined at week 6 using an 8-repetition maximum (8RM) test. Every 4 weeks, the 8RM test is repeated and the cycle repeats.
  Interventions: Behavioral: Aerobic Training; Behavioral: Resistance Training
- Aerobic Training (AT) (Experimental): The AT program will be a four-times-per week program. Twice a week will be AT with a series of standardized AT exercise stations (e.g., treadmills, stationary cycles, aerobic steppers, agility ladders). Participants rotate through each station within the 40-min training duration with approx. 1-min rest between stations. Participants will exercise initially at approximately 50% of their age specific target heart rate reserve and gradually progress to reach the target of 80% of HRR. The other two days per week will be a balance and tone (CON) program consisting of stretching exercises, range of motion exercises, basic core-strength/kegal exercises, static balance exrecises, functional strength exercises (e.g., sit to stand), and relaxation techniques. Other than bodyweight, no additional loading (e.g., hand weights, resistance bands, etc.) will be applied to any of the CON exercises.
  Interventions: Behavioral: Aerobic Training; Behavioral: Balance and Tone Training
- Resistance Training (RT) (Experimental): The RT program will be a four-times-per week program. Twice a week will be RT in which a pressurized air system and free weights will be used to provide the training stimulus. The initial intensity of the training stimulus will be set to a weight where participants can complete 2 sets of 10-15 repetitions. Training intensity will then progress on a cyclic basis from 45 to 85% of predicted 1 RM as determined at week 6 using an 8RM test. Every 4 weeks, the 8RM test is repeated and the cycle repeats.The other two days per week will be a CON program consisting of stretching exercises, range of motion exercises, basic core-strength/kegal exercises, static balance exrecises, functional strength exercises (e.g., sit to stand), and relaxation techniques. Other than bodyweight, no additional loading (e.g., hand weights, resistance bands, etc.) will be applied to any of the CON exercises.
  Interventions: Behavioral: Resistance Training; Behavioral: Balance and Tone Training
- Balance and Tone Program (CON) (Active Comparator): The CON program will be a four-times-per week program. The CON group will consiste of stretching exercises, range of motion exercises, basic core-strength/kegal exercises, static balance exrecises, functional strength exercises (e.g., sit to stand), and relaxation techniques. Other than bodyweight, no additional loading (e.g., hand weights, resistance bands, etc.) will be applied to any of the CON exercises.
  Interventions: Behavioral: Balance and Tone Training

INTERVENTIONS:
Behavioral: Aerobic Training — Six months of twice-weekly aerobic training that will gradually progress in intensity. Each training session will be 60 minutes (10 minutes of warm-up, 40 minutes of training, and 10 minutes of cool-down).
  To meet the public health mandates of COVID-19, when it is necessary, training will occur at home, with the use of wearables to monitor heart rate. Participants will be provided access to instructional videos either by YouTube or DVD. They will be called on a weekly basis to monitor progress and adherence.
  Arms: Aerobic Training (AT); Aerobic Training and Resistance Training (AT&RT)
Behavioral: Resistance Training — Six months of twice-weekly resistance training program that will gradually progress in intensity. Each training session will be 60 minutes (10 minutes of warm-up, 40 minutes of training, and 10 minutes of cool-down).
  To meet the public health mandates of COVID-19, when it is necessary, training will occur at home, with the use of a set of resistance bands of various weights. Participants will be provided access to instructional videos either by YouTube or DVD. They will be called on a weekly basis to monitor progress and adherence.
  Arms: Aerobic Training and Resistance Training (AT&RT); Resistance Training (RT)
Behavioral: Balance and Tone Training — Six months of twice-weekly stretching and relaxation program that includes stretching exercises, range of motion exercises, basic core-strength/kegal exercises, static balance exrecises, functional strength exercises (e.g., sit to stand), and relaxation techniques. Each session will be 60 minutes.
  To meet the public health mandates of COVID-19, when it is necessary, training will occur at home, with the use of small equipment (e.g., pilate ball). Participants will be provided access to instructional videos either by YouTube or DVD. They will be called on a weekly basis to monitor progress and adherence.
  Arms: Aerobic Training (AT); Balance and Tone Program (CON); Resistance Training (RT)
Behavioral: Balance and Tone Training — Six months of twice-weekly stretching and relaxation program that includes stretching exercises, range of motion exercises, basic core-strength/kegal exercises, static balance exrecises, functional strength exercises (e.g., sit to stand), and relaxation techniques. Each session will be 60 minutes.
  To meet the public health mandates of COVID-19, when it is necessary, training will occur at home, with the use of small equipment (e.g., pilate ball). Participants will be provided access to instructional videos either by YouTube or DVD. They will be called on a weekly basis to monitor progress and adherence.
  Arms: Balance and Tone Program (CON)

SUMMARY:
Dementia is one of the most pressing health care issues of the 21st century. Evidence suggests that exercise enhances cognitive function in healthy older adults. Most research has focused on aerobic training (AT). Therefore, investigators aim to assess the individual effects of AT and resistance training (RT), as well as the interaction effect of combining the two types of exercise training, on cognitive function in older adults with mild cognitive impairment.

DETAILED DESCRIPTION:
Investigators will conduct a 6-month assessor-blinded randomized-controlled trial of 216 community-dwelling adults with mild cognitive impairment. Individuals will be randomized to one of four experimental groups, all which receive 6 months of exercise classes four times per week: 1) combined aerobic training and resistance training; 2) aerobic training; 3) resistance training; or 4) balance and toning exercise. There will be two measurement sessions: baseline and 6 months (end of intervention period). A 12-month followup (i.e., 18 months from baseline) measurement will also be done.

ELIGIBILITY:
Inclusion Criteria:

* Community-dwelling in Metro Vancouver
* Have subjective memory complaints, defined as the self-reported feeling of memory worsening with an onset within the last 5 years, as determined by interview and corroborated by an informant
* Have a baseline Montreal Cognitive Assessment (MoCA) score < 26/30
* Mini-Mental State Examination (MMSE) score = or > 22 at screening
* Read, write, and speak English
* Not expected to start or are stable on a fixed dose of anti-dementia medications (e.g., donepezil, galantamine, etc.) during the 6-month intervention period
* Able to walk independently
* Must be in sufficient health to participate in the exercise programs
* Able to comply with scheduled visits, treatment plan, and other trial procedures
* Provide a personally signed and dated informed consent document indicating that the individual (or a legally acceptable representative) has been informed of all pertinent aspects of the trial. In addition, an assent form will be provided at baseline and again at regular intervals

Exclusion Criteria:

* Engaged in moderate (e.g., brisk walking) physical activity > 1 time per week, or > 60 minutes per week, in the 3 months prior to study entry
* Diagnosed with dementia of any type
* Clinically suspected to have neurodegenerative disease as the cause of mild cognitive impairment (MCI) that is not Alzheimer's Disease (AD), vascular cognitive impairment (VCI), or both (e.g., multiple sclerosis, Parkinson's disease, Huntington's disease, frontotemporal dementia)
* At high risk for cardiac complications during exercise or unable to self-regulate activity or to understand recommended activity level; 5) have clinically important peripheral neuropathy or severe musculoskeletal or joint disease that impairs mobility, as determined by his/her family physician
* Taking medications that may negatively affect cognitive function, such as anticholinergics, including agents with pronounced anticholinergic properties (e.g., amitriptyline), major tranquilizers (i.e., typical and atypical antipsychotics), and anticonvulsants (e.g., gabapentin, valproic acid)
* On any hormone therapy (estrogen, progesterone, or testosterone) in the last 24 months
* Planning to participate, or already enrolled in, a concurrent clinical drug or exercise trial

Ages: 65 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 226 (Actual)
Dates: Start 2017-11-13 (Actual); Primary Completion 2024-08-22 (Actual); Study Completion 2025-08-26 (Actual)

PRIMARY OUTCOMES:
Cognitive function as measured by Alzheimer's Disease Assessment Scale Cognitive Subscale Plus (ADAS-Plus) | Baseline to 6 months
  Cognition

SECONDARY OUTCOMES:
Executive functions as measured by standard neuropsychological and computerized tests | Baseline and 6 months and 18 months
  Executive functions
Cardiometabolic risk factors as measured by blood panel | Baseline and 6 months
  Cardiometabolic risk factors
Health related quality of life as measured by the EuroQol five dimensions questionnaire (EQ-5D-5L) | Baseline, 3 months, 6 months, 12 months, and 18 months
  Quality of life
Health related quality of life as measured by the ICE-CAP | Baseline, 3 months, 6 months, 12 months, and 18 months
  Quality of life
Mood as measured by the Center for Epidemiologic Studies Depression Scale (CES-D) | Baseline and 6 months
  Depressive symptoms
Brain function as measured by functional magnetic resonance imaging (fMRI) | Baseline and 6 months
  Brain function
Brain structure as measured by structural magnetic resonance imaging | Baseline and 6 months
  Brain structure
White matter lesion volume as measured by magnetic resonance imaging | Baseline and 6 months
  White matter lesion
Diffusion tensor imaging as measured by magnetic resonance imaging | Baseline and 6 months
  White matter integrity
Memory as measured by standard neuropsychological and computerized tests | Baseline and 6 months and 18 months
  Memory
Visualspatial ability as measured by standard neuropsychological and computerized tests | Baseline and 6 months
  Visualspatial ability
Cardiorespiratory capacity as measured by treadmill test | Baseline and 6 months
  Cardiovascular fitness
Mobility as measured by 400-m walk | Baseline and 6 months and 18 months
  Mobility
Cardiorespiratory capacity esimated from 400-m walk | Baseline and 6 months and 18 months
  Estimated cardiovascular fitness
Cardiometabolic risk as measured by waist to hip ratio | Baseline and 6 months and 18 months
  Cardiometabolic risk
Cardiometabolic risk as measured by body mass index | Baseline and 6 months and 18 months.
  Cardiometabolic risk
Cardiometabolic risk as measured by pulse wave velocity (arterial stiffness) | Baseline and 6 months
  Cardiometabolic risk
Cortisol levels through saliva samples (subset) | 5 times from baseline to 6 months
  Cortisol levels
Lower body strength as measured by the 30 sec sit-to-stand (subset) | Baseline and 6 months and 18 months
  Lower body strength
Lower body strength as measured by Biodex | Baseline and 6 months
  Lower body strength
Upper body strength as measured by grip strength | Baseline and 6 months
  Upper body strength
Sleep quality as measured by Motion Watch actigraphy | Baseline and 6 months
  Sleep quality
Neurotrophic factors as measured by blood | Baseline and 6 months
  Neurotrophic factors
Mobility as measured by Short Physical Performance Battery | Baseline and 6 months and 18 months
  Mobility
Community mobility as measured by the Life Space Questionnaire | Baseline, 3 months, 6 months, 12 months, and 18 months
  Mobility
Body composition as measured by DXA | Baseline and 6 months
  Body composition
Loneliness as measured by the UCLA Loneliness Scale | Baseline and 6 months
  Loneliness
Cognitive function as measured by Alzheimer's Disease Assessment Scale Cognitive Subscale - 13 items | Baseline and 6 months and 18 months
  Cognitive function
Sedentary behaviour as measure by the Sedentary Behaviour Questionnaire | Baseline, 3 months, 6 months, 12 months, and 18 months
  Sedentary behaviour
Risk of sleep apnea as measured by the STOP Bang Questionnaire | Baseline and 6 months
  Sleep apnea risk
Prospective falls via Monthly Calendars | Baseline and 3 months and 6 months and monthly
  Accidental falls
Social support as measured by Social Provision Scale | Baseline and 6 months
  Social support
Mindfulness as measured by the Mindfulness Attention Awareness Scale | Baseline and 6 months
  Mindfulness
Memory as measured by the Everyday Memory Questionnaire | Baseline and 6 months
  Memory
Sleep as measured by the Pittsburgh Sleep Quality Index | Baseline, 6 months, 12 months, and 18 months
  Sleep
Functional ability as measured by the Lawson IADL | Baseline and 6 months
  Instrumental activities of daily living
Comorbidities as measured by the Function Comorbidity Index | Baseline, 6 months, 12 months, and 18 months
  Chronic conditions
Mood as measured by the State and Trait Anxiety Inventory | Baseline and 6 months and 18 months
  Mood
Social network as measured by Lubben Social Network Scale | Baseline and 6 months
  Social network
Physical activity as measured by the CHAMP Questionnaire | Baseline and 3 months and 6 months and monthly
  Physical Activity Level
ADAS-Cog Plus | 18 months
  Cognitive function
Verbal memory and learning using the Rey Auditory Verbal Learning Test | Baseline, 6 months, and 18 months
  Verbal memory and learning
Verbal fluency (categorial of animals and semantic using F,A,S) | Baseline, 6 months, and 18 months
  Verbal functioning tests requiring retrieval
Cytokines - proteins involved in immune response, as measured by blood | Baseline and 6 months
  Cytokines
Dual-task gait using Gaitrite | Baseline and 6 months
  Dual-task walking
Health resource utilization (e.g., access health system services/resources) | Baseline, 3 months, and 6 months
  Access health system services/resources
Physical activity level (i.e., amount of light, moderate, and vigorous) measured by Motion Watch actigraphy | Baseline and 6 months
  Physical activity levels
Sedentary behaviour (i.e., less than = or less than1.5 mets of activity) measured by Motion Watch actigraphy | Baseline and 6 months
  Sedentary behaviour
Quality of life measured by EQ-5D-5L | Baseline, 3 months, 6 months, and 18 months
  Quality of life
Wellbeing measured by ICE-CAP | Baseline, 3 months, 6 months, and 18 months
  Wellbeing
Telemere length | Baseline and 6 months
  Marker of aging
Gait speed over 4-m walk | Baseline, 6 months, and 18 months
  Gait Speed

CONTACTS AND LOCATIONS:
Overall Officials: Teresa Liu-Ambrose, PhD, PT, Principal Investigator — University of British Columbia; John Best, PhD, Principal Investigator — University of British Columbia; Jennifer Davis, PhD, Principal Investigator — University of British Columbia; Lara Boyd, PhD, Principal Investigator — University of British Columbia; Liisa Galea, PhD, Principal Investigator — University of British Columbia; Charlie Goldsmith, PhD, Principal Investigator — Simon Fraser University; Ging-Yuek Robin Hsiung, MD, PhD, Principal Investigator — University of British Columbia; Alexander MacKay, PhD, Principal Investigator — University of British Columbia; Lindsay Nagamatsu, PhD, Principal Investigator — Western University; Claudia Jacova, PhD, Principal Investigator — Pacific University; Arthur Kramer, PhD, Principal Investigator — Northeastern University; Michelle Voss, PhD, Principal Investigator — University of Iowa; Cindy Barha, PhD, Principal Investigator — University of British Columbia; Joel Singer, PhD, Principal Investigator — University of British Columbia
Locations (1):
- University of British Columbia, Vancouver, British Columbia, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Balbim GM, Boa Sorte Silva NC, Falck RS, Kramer AF, Voss MW, Liu-Ambrose T. 24-hour activity cycle behaviors and gray matter volume in mild cognitive impairment. Alzheimers Dement. 2025 Jul;21(7):e70496. doi: 10.1002/alz.70496. PMID 40693459
- [Derived] Barha CK, Falck RS, Best JR, Nagamatsu LS, Hsiung GR, Sheel AW, Hsu CL, Kramer AF, Voss MW, Erickson KI, Davis JC, Shoemaker JK, Boyd L, Crockett RA, Ten Brinke L, Bherer L, Singer J, Galea LAM, Jacova C, Bullock A, Grant S, Liu-Ambrose T. Reshaping the path of mild cognitive impairment by refining exercise prescription: a study protocol of a randomized controlled trial to understand the "what," "for whom," and "how" of exercise to promote cognitive function. Trials. 2022 Sep 9;23(1):766. doi: 10.1186/s13063-022-06699-7. PMID 36085237